CLINICAL TRIAL: NCT04010773
Title: Project for the Liberation of Organizations in an University Hospital in France: A Randomized Controlled Study of the Impact at Two Years of an Intervention Program on the Empowerment of the Medical and Nursing Teams
Brief Title: Impact at Two Years of an Intervention Program on the Empowerment of Medical and Nursing Teams in a French Hospital
Acronym: CHRYSALIDE
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0014
Record Dates: First submitted 2019-06-27; First posted 2019-07-08 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2019-06

CONDITIONS: Empowerment
Keywords: Empowerment; leadership; intervention; psycho-social intervention; motivation; working conditions; occupational health
MeSH Terms: conditions — Empowerment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: collective and psycho-social intervention — The intervention duration is 1 year. It combine (1) In each unit, working groups aimed at improving QWL, (2) counseling and training of directors and frontline managers, and (3) in each unit, concertation meeting between workers, front-line managers and directors.

SUMMARY:
Health in France asks public hospitals to promote quality of working life (QWL), seen as a performance factor. Consistently with empowerment literature, they define QWL as giving workers mastery over their working life. The problem is, French hospitals follow a bureaucratic model, defined by a managerial culture of control and a stratified organization, which weakens mastery of their work, and hinders their commitment and performance. Main objective of CHRYSALIDE, is to create a managerial and organizational transition program of 1 year, and to test its effect at two years on workers empowerment in an university hospital Sub-Center (SC), in comparison with another SC from the same University Hospital Center (CHU) in a randomized controlled study design.

DETAILED DESCRIPTION:
The main objective of CHRYSALIDE is to implement an easy-to-replicate intervention program of 1 year, in order to promote empowering behaviors in directors and front line supervisors in SC, and to test its impact at two years on workers scores of structural empowerment, in comparison with another SC from the same University Hospital Center (CHU).

The secondary objective is to assess the effect of the intervention on psychological empowerment.

To answer to the main objective, quantitative data will be collected three times during the project: Before the implementation, directly after the intervention, and 1 year after the end of the intervention, or 2 years after the beginning. To improve our understanding of what happened during the intervention, a systematic ethnographic report will be done by the investigators and the facilitators engaged in the intervention.

Quantitative data collection will occur during the occupational health visit that is required to be done every two years considering French legislation. For the need of the study, visits will be done every years, and scheduled to match with the beginning and the end of the intervention.

Quantitative data consist in (1) self-reported questionnaires, (2) standardized assessment by medical practitioner during the visit, (3) institutional indicators routinely collected by the SC.

ELIGIBILITY:
Inclusion Criteria:

* Working in one of the care units of the SC that has been randomly selected to benefit from the intervention.

Exclusion Criteria:

Criteria for not including UHPs

* Capacity-building or major reorganization planned during the study period. Criteria for not including services
* Chiefdom of the service opposed to the intervention.
* Strike movement in the team during the inclusion phase. Criteria for not including professionals
* Refusal to participate in the study.
* Physical or psychological condition that prevents the completion of questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all professionals working in the care services of the experimental and control UPHs.
Sampling Method: Non-Probability Sample
Enrollment: 1191 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Structural empowerment, assessed with the Conditions for Work Effectiveness Questionnaire II (CWEQII). | 12 months and 24 months after initial measure.
  This self-reported questionnaire is composed of 19 items about how the worker perceives his work environment. They allow calculation of 6 sub-scores and 1 global score of structural empowerment, reflecting access to the aspects of work environment known to mediate the control of workers over their job. The subscores are "formal power", "informal power", "opportunity", "information", "support" and "resources". They are calculated by summing their specific items, and dividing by 3, except for "informal power" for which the sum is divided by 4. Every sub-score is between 1 and 5. The global score of structural empowerment is calculated by summing the 6 sub-scores. The global score is between 5 and 30. There is not any threshold for the sub-scores and the global score: the higher the scores, the more empowering the working conditions are. The global score is the primary outcome in this study. Safety issue : No.

SECONDARY OUTCOMES:
Psychological empowerment, assessed with the Psychological Empowerment Scale (PES). | 12 months and 24 months after initial measure.
  This self-reported questionnaire is composed of 12 items. They allow calculation of 4 sub-scores and 1 global score of psychological empowerment, reflecting cognitions-believes people with power have about themselves. The sub-scores are "autonomy", "impact", "competence" and "meaning". The sub-scores are calculated by summing their specific items. They are between 15 and 25. The global score is calculated by summing the sub-scores and dividing by 4. It is between 15 and 25. There is not any threshold for the global and sub-scores: the higher the scores, the more people are psychologically empowered. The global score of psychological empowerment is considered as a secondary outcome in this study.
  Safety Issue: No

CONTACTS AND LOCATIONS:
Overall Officials: Baptiste Cougot, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France

REFERENCES:
- [Derived] Cougot B, Gillet N, Moret L, Gauvin J, Caillet P, Fleury-Bahi G, Lesot J, Ollierou F, Armant A, Peltier A, Fouquereau E, Getz I, Bach-Ngohou K, Tripodi D. Relationship between Empowering Leadership and Stress in a French University Hospital: A Cross-Sectional Study Combining the Measurement of Perceived Stress and Salivary Cortisol. J Nurs Manag. 2024 Jan 31;2024:8839893. doi: 10.1155/2024/8839893. eCollection 2024. PMID 40224754
- [Derived] Cougot B, Gillet N, Morin AJS, Gauvin J, Ollierou F, Moret L, Tripodi D. A longitudinal investigation of structural empowerment profiles among healthcare employees. J Nurs Scholarsh. 2024 May;56(3):417-429. doi: 10.1111/jnu.12950. Epub 2023 Dec 13. PMID 38093467
- [Derived] Cougot B, Gillet N, Gauvin J, Caillet P, Fleury-Bahi G, Ollierou F, Armant A, Peltier A, Getz I, Bach-Ngohou K, Tripodi D, Moret L. Impact of empowering leadership on emotional exhaustion: A controlled interventional study in a large French university hospital complex. J Nurs Manag. 2022 Nov;30(8):4234-4250. doi: 10.1111/jonm.13829. Epub 2022 Oct 17. PMID 36190480
- [Derived] Cougot B, Gauvin J, Gillet N, Bach-Ngohou K, Lesot J, Getz I, Deparis X, Longuenesse C, Armant A, Bataille E, Leclere B, Fleury-Bahi G, Moret L, Tripodi D. Impact at two years of an intervention on empowerment among medical care teams: study protocol of a randomised controlled trial in a large French university hospital. BMC Health Serv Res. 2019 Dec 3;19(1):927. doi: 10.1186/s12913-019-4724-7. PMID 31796029